CLINICAL TRIAL: NCT02590601
Title: Bromocriptine in the Treatment of Peripartum Cardiomyopathy, A Bayesian Randomized Registry Trial
Brief Title: Bromocriptine in the Treatment of Peripartum Cardiomyopathy
Acronym: BRO-HF
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not enough patients
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Cardiovascular Society (Other)
Responsible Party: Principal Investigator, Marc Jolicoeur, Lead investigator, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-33-2015-1874 (MP)
Record Dates: First submitted 2015-10-12; First posted 2015-10-29 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Peripartum Cardiomyopathy
Keywords: PPCM; Bromocriptine; Peripartum cardiomyopathy
MeSH Terms: conditions — Peripartum Cardiomyopathy | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bromocriptine + Guideline-driven medical therapy (Active Comparator): In addition to heart failure treatment described above, patients will be administered bromocriptine 2.5 mg orally twice daily for 14 days, followed by 2.5 mg orally daily for 42 days.
  Although not a study procedure, we recommend anticoagulation with prophylactic doses of subcutaneous low-molecular weight heparin during the whole duration of bromocriptine therapy.
  Interventions: Drug: Bromocriptine; Other: Guideline-driven medical therapy (GDMT)
- Guideline-driven medical therapy (Other): New onset PPCM will be managed according to the principles of guideline-driven medical therapy for new-onset heart failure as per the position statement for treatment of PPCM published by the European Society of Cardiology (ESC) and the Canadian Cardiovascular Society (CCS) update on heart failure and pregnancy . The choices and administration of GDMT will be left at the discretion of the treating physician
  Interventions: Other: Guideline-driven medical therapy (GDMT)

INTERVENTIONS:
Drug: Bromocriptine
  Arms: Bromocriptine + Guideline-driven medical therapy
Other: Guideline-driven medical therapy (GDMT)

SUMMARY:
Peripartum cardiomyopathy (PPCM) is a rare, but significant heart disease affecting young women in the puerperal period. Thus far, no specific treatment has been approved to treat this disease. PPCM has a wide spectrum of clinical manifestations ranging from mild heart failure to severe cardiomyopathy, cardiogenic shock and death. A significant proportion of survivors have persistent chronic heart failure leading to disabling symptoms and decreased quality of life.

Animal studies have suggested that prolactin is central to the development of PPCM. Prolactin has pro-inflammatory and anti-angiogenic effects that may promote PPCM. Bromocriptine, a central dopamine agonist known to decrease prolactin levels, might thwart its deleterious effects in women suffering from PPCM. Following this rationale, bromocriptine should improve myocardial function in women suffering from PPCM and thus, improve cardiovascular outcomes and healthcare outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Peripartum cardiomyopathy defined by the following criteria:

   * Development of heart failure in the last month of pregnancy or within 5 months of delivery;
   * Absence of an identifiable alternative cause of heart failure;
   * Absence of recognizable heart disease prior to the last month of pregnancy;
   * Left ventricular systolic dysfunction demonstrated by classic echocardiographic criteria, such as depressed ejection fraction;
3. Recent onset of PPCM ( 1 month);
4. Written informed consent.

Exclusion Criteria:

1. Hypersensitivity or contraindication to bromocriptine;
2. Patients already taking bromocriptine for PPCM or for another indication;
3. Cardiogenic shock before enrolment;
4. Survival expected to be less than 1 year due to non-cardiovascular causes (eg. cancer);
5. Participation to another investigational drug or investigational device study within 30 days prior to randomization (participation to registries is allowed);
6. Patients who in the opinion of the investigator will not comply with specified drugs, or follow-up evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
MACE | 1 year
  MACE : A compose of death from cardiovascular causes, aborted sudden death, heart transplantation, mechanical circulatory support or hospitalization for cardiovascular causes.

SECONDARY OUTCOMES:
Death from cardiovascular causes | 5 years
Left ventricular ejection fraction (LVEF) recovery | 6 months
  Recovery defined as : (proportion of patients with LVEF ≥ 54%)
All-cause mortality | 5 years
Occurence of arrythmias | 1 year
  Arrhythmia : Number of participants with sustained ventricular tachycardia, ventricular fibrillation or new onset atrial fibrillation
Number of all-cause hospitalisation | 5 years
Health-related quality of life (HRQoL) with the Kansas City Cardiomyopathy questionnaire (KCCQ) | 1 year
Health-related quality of life (HRQoL) with the World Health Organization (WHO) quality of life questionnaire (WHOQOL-BREF) | 1 year
Heart transplantation | 5 years
Mechanical circulatory support | 1 year
Number of hospitalisation for cardiovascular causes | 5 years

OTHER OUTCOMES:
Safety adverse events | 12 months
  Safety adverse events: Combined occurence of venous thromboembolic disease, cardiac thrombus with embolic manifestation, myocardial infarction or cerebrovascular accident.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Avram, MD, Principal Investigator — Université de Montréal; Maxime Tremblay-Gravel, MD, MSc, Principal Investigator — Université de Montréal; Guillaume Marquis-Gravel, MD, MSc, Principal Investigator — Université de Montréal; Olivier Desplantie, MD CM, FRCPC, Principal Investigator — Université de Montréal; Anique Ducharme, MD FRCPC, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Monteal, Quebec, Canada

REFERENCES:
- [Derived] Azibani F, Sliwa K. Peripartum Cardiomyopathy: an Update. Curr Heart Fail Rep. 2018 Oct;15(5):297-306. doi: 10.1007/s11897-018-0404-x. PMID 30051292